CLINICAL TRIAL: NCT06425029
Title: SONATA: Self-administered ONe-of-a Kind Approach to Epilepsy Therapy Through a Web-based Music Application
Brief Title: Self-administered ONe-of-a Kind Approach to Epilepsy Therapy Through a Web-based Music Application
Acronym: SONATA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Brian Fidali, MD, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY02002411
Record Dates: First submitted 2024-05-09; First posted 2024-05-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy; Refractory Epilepsy; Music
Keywords: music; epilepsy; responsive neurostimulation; interictal discharge
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: The primary endpoint is to assess the reduction in epileptiform activity (as defined by change in normalized RNS 'long episode' detection frequency) during the 14-day stimulus presentation block for three music pieces. 1) Music piece (A) previously shown to reduce interictal epileptiform discharges (IEDs)). 2) Music piece (B) (previously shown to not reduce IEDs in the same population despite rhythmic similarities), and 3) Music piece (C) - a selection from the participant's preferred musical style that is also matched for musical characteristics.
Who Masked: Participant, Investigator
Masking Description: Participants will not be informed of their group assignment. The study team will have no knowledge of randomization sequence until all participants complete the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Piece A (Experimental): Participants will be asked to listen to a musical excerpt previously shown to have a positive effect on epileptic activity in human brain.
  Interventions: Other: Experimental Intervention (Music A)
- Music Piece B (Active Comparator): Participants will be asked to listen to a musical except very similar to the experimental stimuli that has not been shown to have a positive effect on epileptic activity.
  Interventions: Other: Active Comparator Intervention (Music B)
- Music Piece C (Active Comparator): Participants will select a preferred excerpt from several popular musical genres. This piece is modified to have some similarities to the experimental musical excerpt.
  Interventions: Other: Active Comparator Intervention (Music C)

INTERVENTIONS:
Other: Experimental Intervention (Music A) — Participants will be asked to listen to Music A on their personal device daily, at a time most convenient for them.
  Arms: Music Piece A
Other: Active Comparator Intervention (Music B) — Participants will be asked to listen to music B on their personal device daily, at a time most convenient for them.
  Arms: Music Piece B
Other: Active Comparator Intervention (Music C) — Participants will be asked to listen to music C on their personal device daily, at a time most convenient for them.
  Arms: Music Piece C

SUMMARY:
This is a prospective, placebo-controlled, double-blinded randomized study of self-administered auditory intervention in a naturalistic home environment.

DETAILED DESCRIPTION:
This study aims to replicate and extend findings from prior electrophysiological studies that demonstrated a reduction in epileptiform discharges and seizures in patients living with drug-resistant (medications are not effective) epilepsy after listening to specific music.

It is believed to be the first study to examine the effect of daily, self-administered musical stimuli in reduction of epileptiform event detections over days to weeks. The study will enroll a cohort of patients already implanted with NeuroPace Responsive Neurostimulator (RNS) device to treat their epilepsy. This device uses continuous, outpatient electrocorticographic recording data to provide immediate (or 'responsive') closed loop neurostimulation.

Primary hypothesis is that patients with drug resistant epilepsy, implanted with RNS, will have fewer epileptic activity episodes (RNS 'long episodes') during the weeks of experimental music intervention. The study team expect to see improvement with daily listening to specific music intervention (experimental, Music A), but not with active comparators (Music B or C). The effect, if any, of music intervention is expected to last at least one week after the intervention period (block) (for each music piece) ends.

Secondary hypothesis is that the music listening every day will be associated with improved self-report of mood, quality of life, and self-reported measures of cognition. The study team suspects that this effect will not be limited to just one specific musical piece.

This study will also look to determine the feasibility of an at-home, self-administered auditory intervention in drug resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Adults with medication-refractory focal epilepsy who have undergone RNS implantation at least six months prior and are in the judgement of the treating physician on a stable RNS regimen in terms of stimulation
* Willing to attend all study visits and complete all required study procedures
* Access to private or public wireless data service at regular intervals
* Access to personal mobile device

Exclusion Criteria:

* Documentation of a musicogenic, or auditory-triggered focal seizure semiology
* Participant is unable to reasonably participate in study tasks as determined by the investigator
* Inability to obtain informed consent from the patient or legally authorized representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Music Intervention and its effects on epileptic activity in human brain | Baseline, Week 3-4, Week 9-10, and Weeks 13-14, (Approximately 4 1/2 Months)
  This measure aims to determine if specific music intervention has positive effect on epileptic activity in participants with responsive neurostimulation device (RNS) implanted for drug-resistant epilepsy (DRE). The effect will be measured as a change in the number of "long episodes" or epileptic activity in a participants' brain as detected and recorded by the RNS device before and after study music interventions.

SECONDARY OUTCOMES:
Reduction in patient-reported seizures | Throughout the study completion, an average of 5 1/2 months (4 weeks retrospective data collection and 4 1/2 months post enrollment)
  The study team will collect and assess the number of seizures reported by participants during the 4-week period before enrollment (retrospective or going back in time) and 4 1/2 months throughout the study (prospective or going forward in time).
Determining duration of therapeutic effect of music intervention | Throughout the study completion, an average of 5 1/2 months (4 weeks retrospective data collection and 4 1/2 months post enrollment)
  The study team will assess the time frame (seconds, hours, days, weeks, etc.) during which the reduction of "long episodes" or epileptic activity in participants' brain, as detected by the RNS system, lasts after each music intervention.
Assessment of pre- and post-intervention cognition scores (BRIEF-A) | Throughout the study completion, an average of 5 1/2 months (4 weeks retrospective data collection and 4 1/2 months post enrollment)
  The study team will measure this outcome by comparing the difference in individual scores collected via cognition questionnaire (BRIEF-A) done by all participants before study intervention (Enrollment Visit) and at the end of the study ("End of Study" visit).
Assessment of pre- and post-intervention mood (DASS-21) | Throughout the study completion, an average of 5 1/2 months (4 weeks retrospective data collection and 4 1/2 months post enrollment)
  The study team will measure this outcome by comparing the difference in individual scores collected via mood questionnaire (DASS-21) done by all participants before study intervention (Enrollment Visit) and at the end of the study ("End of Study" visit).
Assessment of pre- and post-intervention quality of life (QOLIE-31) | Throughout the study completion, an average of 5 1/2 months (4 weeks retrospective data collection and 4 1/2 months post enrollment)
  The study team will measure this outcome by comparing the difference in individual scores collected via quality-of-life questionnaire (QOLIE-31) done by all participants before study intervention (Enrollment Visit) and at the end of the study ("End of Study" visit).
Assessment of music preferences pre- and post-intervention | Throughout the study completion, an average of 5 1/2 months (4 weeks retrospective data collection and 4 1/2 months post enrollment)
  The study team will review participants' responses to study specific music questionnaire. The outcome will be measured as percentage of participants and their specific musical preferences pre- and post-intervention.
Assess feasibility of real-world, at home auditory stimulus interventions for patients with drug resistant epilepsy | Throughout the study completion, an average of 5 1/2 months (4 weeks retrospective data collection and 4 1/2 months post enrollment)
  The study team will assess participants' engagement with study interventions over the course of this study. This will be measured as a number of days each participant missed each music intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Fidali, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: No
The study results will be available on ClinicalTrials.gov and will be published in appropriate clinical journal upon completion.

REFERENCES:
- [Background] Quon RJ, Casey MA, Camp EJ, Meisenhelter S, Steimel SA, Song Y, Testorf ME, Leslie GA, Bujarski KA, Ettinger AB, Jobst BC. Musical components important for the Mozart K448 effect in epilepsy. Sci Rep. 2021 Sep 16;11(1):16490. doi: 10.1038/s41598-021-95922-7. PMID 34531410
- [Background] Feng Y, Quon RJ, Jobst BC, Casey MA. Evoked responses to note onsets and phrase boundaries in Mozart's K448. Sci Rep. 2022 Jun 10;12(1):9632. doi: 10.1038/s41598-022-13710-3. PMID 35688855